CLINICAL TRIAL: NCT03134937
Title: Does High-Flow Heated and Humidified Nasal Oxygen Therapy (HFHHNO) Result in Gastric Distension? A Two-center Prospective Study
Brief Title: High-Flow Heated and Humidified Oxygen Therapy and Gastric Distension
Acronym: HFHHNOGastric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-5152
Record Dates: First submitted 2017-02-16; First posted 2017-05-01 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-02

CONDITIONS: Gastric Distention
Keywords: Gastric Ultrasound; Gastric Distension; Gastric Volume; Gastric Fluid Volume; High-flow oxygen therapy; HFHHNO; Healthy volunteer

STUDY DESIGN:
Intervention Model Description: Every participant will recieve one HFHHNO session, will get 30 mins of oxygen up to 60-70 L/min.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Other): Participants will undergo one session of high-flow heated and humidified oxygen therapy (HFHHNO) (up to 60-70 litre/min). They will undergo a gastric ultrasound scan after session of HFHHNO therapy.
  Interventions: Device: High-Flow Heated and Humidified Oxygen Therapy (HFHHNO)

INTERVENTIONS:
Device: High-Flow Heated and Humidified Oxygen Therapy (HFHHNO) — Participants will undergo one session of high-flow heated and humidified oxygen therapy (HFHHNO) (up to 60-70 litre/min). They will undergo a gastric ultrasound scan after session of HFHHNO therapy.

SUMMARY:
High Flow Heated and Humidified Nasal Oxygen therapy (HFHHNO) has been increasingly used in emergency medicine to assist patients with short term respiratory failure and to provide adequate oxygen to the body prior to intubation.

Gastric distension which is the bloating of the stomach due to air being pumped into it is a concern for anesthesiologists as it increases the risk of nausea and vomiting during surgery (aspiration).

The objective of this study is use an ultrasound machine to measure the volume of fluid in the stomach before and after HFNO is used in a standard clinical manner.

DETAILED DESCRIPTION:
High Flow Heated and Humidified Nasal Oxygen therapy (HFHHNO) is being increasingly used in the emergency medicine and intensive care settings to manage patients with acute hypoxemic respiratory failure, and to optimize pre-oxygenation prior to intubation in patients with mild-to-moderate hypoxemia.

More recently, there have been reports of applications in the anesthesia perioperative setting. In fact, it is possible that the single greatest potential advantages of HFHHNO for anesthesia practice is that (unlike face mask and CPAP devices) oxygen administration can be maintained during periods of apnea with the potential to significantly prolong the apnea time available for safe and effective airway management.

However, the low levels of positive airway pressure associated with HFHHNO has raised the question of whether prolonged use could result in gastric insufflation thus increasing the risk of regurgitation and aspiration with an unprotected airway. Gastric distension is a concern for anesthesiologists because it leads to the activation of a parasympathetically-mediated reflex through the vagus nerve that leads to secretion of acetylcholine by enteric neurons. In turn, increased acetylcholine activates M3 receptors on parietal cells resulting in increased secretion of gastric acid. The combination of an increased volume of gastric secretions and high intraluminal pressure may place patients at risk of pulmonary aspiration.

The primary objective will be any change in gastric fluid volume from the baseline to each scan following HFHHNO therapy. Participants will undergo an abdominal ultrasound scan prior to any oxygen therapy to provide a baseline. One 30-minute session of oxygen therapy will follow(up to 60-70 L/min). After session, another ultrasound scan will take place, identical to the baseline to obtain the same measurements. From the images taken by the ultrasound, a mathematical model can be applied to calculate the gastric volume (and any change).

The secondary outcome will be the incidence of "gastric air distension" defined by qualitative ultrasound as a distended antrum with air content that blurs the posterior gastric wall.

ELIGIBILITY:
Inclusion Criteria

1. Healthy volunteers aged 18 to 70 years
2. Male or female
3. American Society of Anesthesia physical status classification I and II
4. Height greater than 145 cm
5. Ability to understand the study protocol and provide informed consent. Communication difficulties will not be an impediment to participate. In case of a language barrier, translation services will be sought as per usual institutional practice.

Exclusion Criteria

1. Subjects predisposed to have an increased residual gastric volume at baseline (e.g. diabetes or known gastric dysmotility)
2. History of major upper gastrointestinal disease (including hiatus hernia or prior gastroduodenal surgery)
3. Morbid obesity (Body Mass Index > 40 Kg/m2)
4. Chronic Obstructive Pulmonary Disease (Emphysema or Chronic Bronchitis)
5. Subjects diagnosed with type I and II Diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Change in Gastric Volume | Prior to, and immediately following session of HFHHNO oxygen therapy.
  Ultrasound scan will be used to determine if there was an increase in gastric fluid volume following session of oxygen therapy.

SECONDARY OUTCOMES:
Gastric Distension | Immediately following session of HFHHNO oxygen therapy.
  The secondary outcome will be the incidence of "gastric air distension" defined by qualitative ultrasound as a distended antrum with air content that blurs the posterior gastric wall.

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Perlas, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD is to be shared with other researchers. All data will be obtained during an gastric ultrasound scan.

REFERENCES:
- [Derived] McLellan E, Lam K, Behringer E, Chan V, Bozak D, Mitsakakis N, Perlas A. High-flow nasal oxygen does not increase the volume of gastric secretions during spontaneous ventilation. Br J Anaesth. 2020 Jul;125(1):e75-e80. doi: 10.1016/j.bja.2020.02.023. Epub 2020 Mar 31. PMID 32241548